CLINICAL TRIAL: NCT06507891
Title: A Phase Ib, Open-label, Dose Escalation and Expansion Study to Evaluate the Tolerance , Pharmacokinetics and Effectiveness of TQ-A3334 Tablets in Patients With Advanced Non-small Cell Lung Cancer
Brief Title: A Clinical Study to Evaluate the Tolerance, Pharmacokinetics and Efficacy of TQ-A3334 Tablets
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: After considering the company's project situation and strategic development direction, it has been decided to terminate this project. The experiment will be terminated for non safety reasons.
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQ-A3334-I-02
Record Dates: First submitted 2024-07-11; First posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQ-A3334 tablets (Experimental): TQ-A3334 tablets administered orally on day 1, 8, 15 in 21-day cycle.
  Interventions: Drug: TQ-A3334 tablets
- TQ-A3334 tablets + Anlotinib capsules (Experimental): TQ-A3334 tablets administered orally on day1, 8, 15 in 21-day cycle plus Anlotinib capsules given orally in fasting conditions , once daily in 21-day cycle (14 days on treatment from Day 1-14, 7 days off treatment from Day 15-21).
  Interventions: Drug: TQ-A3334 tablets + Anlotinib capsules

INTERVENTIONS:
Drug: TQ-A3334 tablets — TQ-A3334 is a highly efficient and highly selective Toll-like receptor-7 (TLR-7) agonist. TLR-7 can induce the release of a series of pro-inflammatory cytokines, including interferon alpha (IFN-α), Interleukin 12 (IL-12), Tumor Necrosis Factor Alpha (TNF-α), and promote the maturation and antigen presentation of dendritic cells, play an antitumor effect.
  Arms: TQ-A3334 tablets
Drug: TQ-A3334 tablets + Anlotinib capsules — TQ-A3334 is a highly efficient and highly selective TLR-7 agonist. TLR-7 can induce the release of a series of pro-inflammatory cytokines, including IFN-α (interferon-α), IL-12 (Interleukin 12), TNF-α, and promote the maturation and antigen presentation of dendritic cells, play an antitumor effect.
  Anlotinib hydrochloride is a muti-target tyrosine kinase inhibitor.
  Arms: TQ-A3334 tablets + Anlotinib capsules

SUMMARY:
This is a study to evaluate the tolerance, dose-limiting toxicity (DLT), and maximum tolerated dose (MTD) of single and multiple oral doses of TQ-A3334 and observe the efficacy of TQ-A3334 in combination with anlotinib capsules in patients with non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Understood and signed an informed consent form;
* 18 years old and older; Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 1; life expectancy ≥12 weeks;
* Histologically confirmed advanced non-small cell lung cancer;
* Has received at least two systemic chemotherapy regimens which is failure or intolerance；
* At least one measurable lesion（ based on Response evaluation criteria in solid tumors (RECIST) 1.1;
* The main organs function are normally；
* Male or female subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 6 months after the last dose of study (such as intrauterine devices , contraceptives or condoms) ；No pregnant or breastfeeding women, and a negative pregnancy test are received within 7 days before the randomization；
* In addition to the above criteria, the extended research phase must meet the following criteria: epidermal growth factor receptor (EGFR) and anaplastic lymphoma kinase (ALK) are negative; or patients with positive test results of EGFR and ALK are resistant or intolerant after receiving the targeted drug treatment.

Exclusion Criteria:

* Small cell lung cancer
* Other malignant tumors that have appeared or are presently present within 5 years, except for cured cervical carcinoma in situ and non-melanoma skin cancer
* Has received chemotherapy, surgery, radiotherapy, the last treatment from the first dose less than 4 weeks, or oral targeted drugs for less than 5 half-lives, or oral fluorouracil pyridine drugs for less than 14 days, mitomycin C and nitrosourea for less than 6 weeks
* Expect to use any active vaccine against infectious diseases within 28 days before the first administration or during the study period
* Immunosuppressive therapy with immunosuppressive agents or systemic or absorbable local hormones (dosage > 10 mg/day prednisone or other therapeutic hormones) is required for the purpose of immunosuppression, and is still in use for 2 weeks after the first administration
* Active autoimmune diseases that require systemic treatment have occurred within 2 years before the first administration
* Hypersensitivity to TQ-A3334 or its excipient
* Has uncontrollable symptoms of brain metastases, spinal cord compression, cancerous meningitis
* Has unrelieved toxicity reactions ≥ grade 1 due to previous treatment
* Imaging (CT or MRI) shows that tumor invades large blood vessels or the boundary with blood vessels is unclear
* Has thyroid dysfunction that requires drug treatment within 6 months before the first administration
* Has multiple factors affecting oral medication
* Has any severe acute complications before the first administration
* Have participated in other clinical trials within 4 weeks before the first administration
* According to the judgement of the researchers, there are other factors that may lead to the termination of the study
* In addition to the above criteria, the extended research phase must meet the following criteria:

  1. Pathologically diagnosed as central, hollow lung squamous cell carcinoma, or non-small cell lung cancer with hemoptysis;
  2. EGFR and ALK are positive untreated with relevant targeted drugs;
  3. Has received anlotinib hydrochloride capsules.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2023-08-25 (Actual); Study Completion 2024-06-04 (Actual)

PRIMARY OUTCOMES:
Adverse events (AE) | Baseline up to 21 days
  The occurrence of adverse events and serious adverse events.
Dose limited toxicity (DLT) | Baseline up to 21 days
  DLT defined as any of the following events occurring during the study related to drugs: (1) ≥grade 3 non-hematologic toxicity; (2) Grade 4 neutropenia, thrombocytopenia, and hemoglobin reduction confirmed by at least 2 tests within 2 days; (3) Grade 3 neutropenia with fever confirmed at least 2 times within 2 days; (4) Immune-related interstitial pneumonia ≥ grade 2; (5) Decreased ventricular ejection fraction ≥ grade 2 ; (6) Retinal vein occlusion (RVO), uveitis ≥ grade 2.
Maximum tolerable dose (MTD) | Baseline up to 21 days
  MTD defined as the highest dose level at which less than or equal to 2 of 6 subjects experience dose limiting toxicity (DLT).

SECONDARY OUTCOMES:
Tmax | 5 minutes, 15 minutes, 0.5 hour, 45 minutes, 1 hour, 1.5 hour, 4 hour, 12 hour, 24 hour, 48 hour, 96 hour, 144 hour after oral administration on day 1 and day 29; 30 minutes before oral administration on day 1, day 8, day 15,day 22 and day 29
  To characterize the pharmacokinetics of TQ-A3334 by assessment of time to reach maximum plasma concentration.
Cmax | 5 minutes, 15 minutes, 0.5 hour, 45 minutes, 1 hour, 1.5 hour, 4 hour, 12 hour, 24 hour, 48 hour, 96 hour, 144 hour after oral administration on day 1 and day 29; 30 minutes before oral administration on day 1, day 8, day 15,day 22 and day 29
  Cmax is the maximum plasma concentration of TQ-A3334 or metabolite(s).
t1/2 | 5 minutes, 15 minutes, 0.5 hour, 45 minutes, 1 hour, 1.5 hour, 4 hour, 12 hour, 24 hour, 48 hour, 96 hour, 144 hour after oral administration on day 1 and day 29; 30 minutes before oral administration on day 1, day 8, day 15,day 22 and day 29
  t1/2 is time it takes for the blood concentration of TQ-A3334 or metabolite(s) to drop by half.
Area under the plasma concentration-time curve (AUC 0-t) | 5 minutes, 15 minutes, 0.5 hour, 45 minutes, 1 hour, 1.5 hour, 4 hour, 12 hour, 24 hour, 48 hour, 96 hour, 144 hour after oral administration on day 1 and day 29; 30 minutes before oral administration on day 1, day 8, day 15,day 22 and day 29
  To characterize the pharmacokinetics of TQ-A3334 by assessment of area under the plasma concentration time curve from zero to infinity.
Overall response rate (ORR) | Up to 96 weeks
  Percentage of Participants Achieving Complete Response (CR) and Partial Response (PR).
Progression-free survival (PFS) | Up to 96 weeks
  PFS defined as the time from randomization until the first documented progressive disease (PD) or death from any cause.
Duration of Response (DOR) | Up to 96 weeks
  Time from tumor first assessment to CR or PR to first assessment to PD (Progressive Disease) or death from any cause.
Disease control rate (DCR) | Up to 96 weeks
  Percentage of Participants Achieving Complete Response (CR) and Partial Response (PR) and Stable Disease (SD).

CONTACTS AND LOCATIONS:
Locations (1):
- Jingling Hospital, Nanjing, Jiangsu, China